CLINICAL TRIAL: NCT00365560
Title: A Randomised, Double-Blind, Placebo-Controlled, Crossover Efficacy and Safety Evaluation of 8-Week Treatment Periods of Two Doses [5 Mcg (2 Actuations of 2.5 Mcg) and 10 Mcg (2 Actuations of 5 Mcg)] of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler® as Add-on Therapy in Patients With Severe Persistent Asthma
Brief Title: An Efficacy and Safety Evaluation of Tiotropium add-on Therapy in Patients With Severe Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.341
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium
Drug: placebo

SUMMARY:
The primary objective of this study is to examine efficacy and safety of tiotropium compared to plac ebo as add-on therapy in severe asthmatics according to GINA step 4 classification

ELIGIBILITY:
Inclusion Criteria:

Outpatients of either sex, age 18 - 75 years, with at least a documented 5 year history of asthma, and a current diagnosis of severe, persistent asthma (GINA step 4), smoking history < 10 pack years and >= 1 year smoking cessation; Patients must be symptomatic

Exclusion Criteria:

Patients

* with a recent history (i.e., six months or less) of myocardial infarction,
* who have been hospitalized for heart failure (NYHA class III or IV) within the past year,
* with any unstable or life threatening cardiac arrhythmia or cardiac arrhythmia requiring intervention or a change in drug therapy within the past year,
* with malignancy for which the patient has undergone resection, radiation ther apy or chemotherapy within the last five years,
* who have undergone thoracotomy with pulmonary resection,
* with moderate to severe renal impairment (creatinine clearance = 50 mL/min)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115
Dates: Start 2006-08; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the FEV1 response (within 3 hours post dosing) determined at the end of the 8-week treatment period

SECONDARY OUTCOMES:
FEV1 and FVC AUC 0-3h (in a subset 0-24h) PEF, use of rescue medication, daytime and nocturnal symptoms etc.

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (16):
- Denmark (5):
  - Boehringer Ingelheim Investigational Site, Aalborg
  - Boehringer Ingelheim Investigational Site, Aarhus C
  - Boehringer Ingelheim Investigational Site, Hvidovre
  - Boehringer Ingelheim Investigational Site, K?benhavn NV
  - Boehringer Ingelheim Investigational Site, Odense C
- Germany (5):
  - Boehringer Ingelheim Investigational Site, Gelnhausen
  - Boehringer Ingelheim Investigational Site, Gro?hansdorf
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
  - Boehringer Ingelheim Investigational Site, Wiesbaden
  - Boehringer Ingelheim Investigational Site, Wiesloch
- Netherlands (6):
  - lokatie Langendijk, Breda
  - Polikliniek longziekten, Eindhoven
  - Polikliniek longziekten, Groningen
  - Polikliniek Longziekten, Heerlen
  - Polikliniek longziekten, Hengelo
  - lokatie het Spittaal, Zutphen

REFERENCES:
- [Derived] Kerstjens HA, Disse B, Schroder-Babo W, Bantje TA, Gahlemann M, Sigmund R, Engel M, van Noord JA. Tiotropium improves lung function in patients with severe uncontrolled asthma: a randomized controlled trial. J Allergy Clin Immunol. 2011 Aug;128(2):308-14. doi: 10.1016/j.jaci.2011.04.039. Epub 2011 Jun 2. PMID 21636120